CLINICAL TRIAL: NCT01561183
Title: Vital Pulp Therapy for Management of Irreversible Pulpitis in Human Permanent Teeth: A Randomized Clinical Trial.
Brief Title: Vital Pulp Therapy (VPT) Using Calcium Enriched Mixture (CEM) to Treat Irreversible Pulpitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Saeed Asgary, Dean of ICER, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IKHDC: 01-11-1390
Record Dates: First submitted 2012-03-14; First posted 2012-03-22 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Irreversible Pulpitis
Keywords: Vital pulp therapy; Pulp cap; pulpotomy; calcium enriched mixture; CEM cement; Endodontic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Indirect pulp capping (IPC) (Experimental): Indirect pulp capping
  Interventions: Procedure: Indirect pulp capping (IPC)
- Direct pulp capping (DPC) (Experimental): Direct pulp capping
  Interventions: Procedure: Direct pulp capping (DPC)
- Miniature pulpotomy (MP) (Experimental): Miniature pulpotomy
  Interventions: Procedure: Miniature pulpotomy (MP)
- Full pulpotomy (FP) (Experimental): Full pulpotomy
  Interventions: Procedure: Full pulpotomy (FP)

INTERVENTIONS:
Procedure: Indirect pulp capping (IPC) — Procedure: IPC
  The IPC will be performed as follow:
  * Anesthesia
  * isolation the tooth
  * access to the lesion
  * incomplete removal of carious tissue from the cavity walls
  * indirect pulp capping with ≈2 mm layer calcium enriched mixture cement
  * permanent filling with sandwich technique
  Other Names: Indirect pulp capping
  Arms: Indirect pulp capping (IPC)
Procedure: Direct pulp capping (DPC) — Procedure: DPC
  The DPC will be performed as follow:
  * Anesthesia
  * isolation the tooth
  * access to the lesion
  * complete removal of carious tissue from the cavity walls result in pulp exposure
  * preparation of clot-free pulpal mound
  * direct pulp capping with ≈2 mm layer calcium enriched mixture cement
  * permanent filling with sandwich technique
  Other Names: Direct pulp capping
  Arms: Direct pulp capping (DPC)
Procedure: Miniature pulpotomy (MP) — Procedure: MP
  The MP will be performed as follow:
  * Anesthesia
  * isolation the tooth
  * access to the lesion
  * complete removal of carious tissue from the cavity walls result in pulp exposure
  * intentionally removal of pulp horn (≈1 mm)
  * preparation of clot-free pulpal mound
  * direct pulp capping with ≈2 mm layer calcium enriched mixture cement
  * permanent filling with sandwich technique
  Other Names: Miniature pulpotomy
  Arms: Miniature pulpotomy (MP)
Procedure: Full pulpotomy (FP) — Procedure: FP
  The FP will be performed as follow:
  * Anesthesia
  * isolation the tooth
  * access to the lesion
  * complete removal of carious tissue from the cavity walls result in pulp exposure
  * pulpotomy
  * preparation of clot-free pulpal mound
  * direct pulp capping with ≈2 mm layer calcium enriched mixture cement
  * permanent filling with sandwich technique
  Other Names: Full pulpotomy
  Arms: Full pulpotomy (FP)

SUMMARY:
To compare the effect of different VPT methods using Calcium Enriched Mixture (CEM) cement for management of human dental pulp with irreversible pulpitis.

DETAILED DESCRIPTION:
The purpose of this randomized clinical trial is to demonstrate the effect of four methods of Vital Pulp Therapy (VPT) using a new endodontic bio-material [calcium enriched mixture (CEM) cement] in pain relief as well as clinical/radiographic success, for management of irreversible pulpitis of human permanent teeth.

ELIGIBILITY:
Inclusion Criteria:

1. Carious permanent vital mature molar tooth with closed apex (with preoperative X-ray)
2. Positive response to EPT or cold test
3. patients willing to participate in study
4. Healthy subjects; absence of any systematic disorder
5. Age ≥ 10 years old
6. Both gender
7. Written informed consent

Exclusion Criteria:

1. Moderate or severe periodontitis; pockets >3mm
2. None restorable tooth
3. Internal or external root resorption
4. Root canal calcification
5. Non vital pulps
6. Analgesic taken within the last 8h
7. Active systemic disease
8. Pregnancy or nursing
9. History of opioid addiction/abuse
10. Temporary residency

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2012-03; Primary Completion 2014-03 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Clinical and radiographical success rates (%) of each treatment group | 1 year
  The outcome of clinical success/failure is determined by subjective symptoms and objective observation of inflammation/infection.
  The outcome of radiographic success is classified by using a modification of the Strindberg criteria.

SECONDARY OUTCOMES:
Patient Assessment of Pain with questionnaire | 6-months
  Pain assessment is carried out using the pain Numerical Rating Scale (NRS) with ratings between 0 to 9. Pain assessment is made up to 7 days. One NRS form is given to each patient to complete.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Jafar Eghbal, DDS, MS, Study Director — Iran Center For Dental Research
Locations (1):
- Imam Khomeini Dental Clinic, Tehran, Iran

REFERENCES:
- [Background] Asgary S, Ahmadyar M. Can miniature pulpotomy procedure improve treatment outcomes of direct pulp capping? Med Hypotheses. 2012 Feb;78(2):283-5. doi: 10.1016/j.mehy.2011.11.002. Epub 2011 Dec 1. PMID 22137499